CLINICAL TRIAL: NCT01966094
Title: Observational Study of HIV-associated Neurocognitive Disorder
Acronym: HAND2
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Albert ML Anderson, Principal Investigator, Emory University
Other Study IDs: IRB00065880; K23MH095679 (NIH)
Record Dates: First submitted 2013-09-12; First posted 2013-10-21 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: HIV Associated Neurocognitive Disorder; Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (plasma) samples and cerebrospinal fluid (CSF)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HIV+ subjects with HAND: Human immunodeficiency virus (HIV) positive subjects with HIV-associated neurocognitive disorder (HAND) and either antiretroviral therapy (ART) naïve or ART-experienced off treatment for at least 6 months
- HIV+ subjects without HAND: Human immunodeficiency virus (HIV) positive subjects without HIV-associated neurocognitive disorder (HAND) and either antiretroviral therapy (ART) naïve or ART-experienced off treatment for at least 6 months

SUMMARY:
It is estimated that over 1 million people in the United States have HIV infection. While HIV is treatable, there are still high rates of HIV-associated neurocognitive disorder (HAND). HAND is defined by low scores on memory testing. To meet the criteria for HAND, an HIV-infected individual has to have a low score on at least two different memory tests. It is estimated that 20-50% of people living with HIV have HAND. It is therefore still a common problem. While individuals with HAND typically improve on antiretroviral therapy for HIV, often this improvement is incomplete. Also, there are over 20 antiretroviral medications approved for HIV in the US. It is not clear if the specific choice of antiretroviral medication makes a difference in the improvement of HAND.

The investigators have designed a small preliminary study in which subjects with and without HAND who have never been on treatment for HIV or have been off treatment for at least 6 months are followed for the first 12 months after starting antiretroviral therapy.The investigators will enroll a maximum of 46 subjects (23 subjects in each arm). Subjects will also be followed by their primary HIV medical provider. For the study, subjects will be followed for 48 weeks. There are three followup visits: 12 weeks, 24 weeks, and 48 weeks. Memory testing will be performed at baseline and each followup visit. Blood will also be taken at baseline and the three followup visits to measure changes in inflammation. A lumbar puncture will be performed at baseline and at 24 weeks to measure changes in inflammation and amount of HIV virus in the spinal fluid. There is also an optional lumbar puncture at the last study visit of 48 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV infection (HAART naïve), subjects 18 to 59 years of age
2. Negative serum cryptococcal antigen if CD4+ T-cell count <100 cells/microliter, normal serum thyroid stimulating hormone level, negative serum rapid plasma reagin (RPR) (Can have positive RPR ≤1:4 if treated for syphilis by CDC guidelines at least 6 months prior to enrollment, had no signs/symptoms of neurosyphilis, and RPR titer decreased at least 4-fold by 6 months after treatment).

Exclusion Criteria:

1. Ongoing heavy alcohol use (more than 2 drinks per day) or ongoing illicit drug use
2. Schizophrenia or other psychotic disorder, bipolar disorder, or uncontrolled depression as reported by the subject or medical provider.

3 Neoplasm of the CNS OR history of traumatic brain injury with loss of consciousness > 30 minutes OR CNS infection in the last 6 months.

4. Pregnancy or incarceration

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects will be identified through referrals from HIV medical providers in the Atlanta metropolitan area. Potential subjects will be recruited from the Grady Infectious Diseases clinic as well as other clinics in the metropolitan Atlanta area, which include the Fulton and Dekalb county health departments, the Emory Infectious Diseases clinic, as well as private HIV medical practices in the area.
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2013-10; Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Difference in neurocognition change over 48 weeks as measured by a summary score (NPZ-8) that reflects an 8 test neurocognitive battery. | 48 weeks
  NPZ-8 scores will be determined at each of the four visits (baseline, 12 weeks, 24 weeks, and 48 weeks). The NPZ-8 score equals the subject score minus the mean age adjusted score divided by the standard deviation of the second score.

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States